CLINICAL TRIAL: NCT01312480
Title: Adolescent Smoking Cessation in Pediatric Primary Care
Acronym: Smokebusters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Academy of Pediatrics (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jonathan D. Klein, Professor of Pediatrics, University of Illinois at Chicago, American Academy of Pediatrics
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SB-1R01CA140576-01A2; 1R01CA140576-01A2 (NIH)
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Tobacco Cessation; Media Use
Keywords: Tobacco; Tobacco Prevention; Tobacco Cessation; 5A's Model; Adolescence; Media Use
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Other): The smoking cessation intervention is a Public Health Services-approved intervention based on the 5A's Model, which includes (1) Ask if the patient smokes, (2) Advise every patient to quit, (3) Assess readiness to quit, (4) Assist in quitting and finding services and (5) Arrange for cessation services and follow up. Practitioners will complete a 5A checklist for each patient in this arm.
  Interventions: Other: 5A's Model
- Control Group (Other): The media use assessment (control condition) is based in part on the American Academy of Pediatrics policy statement on children and media, published in the November 2010 issue of Pediatrics. This assessment includes suggested questions on how much media per day is used and whether or not the adolescent has a television or Internet access in his/her bedroom. The adolescent will complete a one-page Media Use assessment form for this purpose, which will set the stage for relevant anticipatory guidance.
  Interventions: Other: Media Use Assessment

INTERVENTIONS:
Other: 5A's Model — The smoking cessation intervention is based on the 5A's model, which includes the following elements:
  1. Ask if the patient smokes.
  2. Advise every patient to quit.
  3. Assess readiness to quit.
  4. Assist in quitting and finding services.
  5. Arrange for cessation services and follow-up.
  Arms: Intervention Group
Other: Media Use Assessment — The media use assessment (control condition) is based in part on the American Academy of Pediatrics policy statement on children and media, published in the November 2010 issue of Pediatrics. This assessment includes suggested questions on how much media per day is used and whether or not the adolescent has a television or Internet access in his/her bedroom. The adolescent will complete a one-page Media Use assessment form for this purpose, which will set the stage for relevant anticipatory guidance.
  Arms: Control Group

SUMMARY:
This is a study of the effectiveness of adolescent smoking cessation interventions in pediatric primary care settings. Our specific aims are to:

1. Demonstrate providers' fidelity to guidelines for tobacco counseling and delivery of cessation interventions using practice system changes over time, (including systematic screening using charting tools and linkages to adjunct materials, including self-help handouts and Internet resources); and
2. Assess the impact of primary care provider counseling interventions on adolescent smoking cessation.

We hypothesize that adolescents who receive guidelines-based clinician-delivered smoking cessation counseling at primary care visits will be more likely to make quit attempts and more likely to remain abstinent (with better long term cessation rates) at 6 and 12 months after intervention, compared to those who do not receive interventions. In addition, we hypothesize that successful referral to stage-based self-help adjuncts, and more adjunct use will be associated with more quit attempts and better long-term cessation rates.

We will evaluate provider interventions in up to 120 pediatric practices, recruited from the American Academy of Pediatric's Pediatric Research in Office Settings (PROS) practice-based research network. Adolescents presenting for care will complete a short baseline survey prior to their doctor-visit, and a percentage of participants will be surveyed by phone 4-6 weeks after their visits to assess quit attempts and short-term cessation, and again at 6 and 12 months to evaluate long-term cessation outcomes. We will describe the patterns of smoking among youth, and explore how much receiving interventions affects motivation, quitting, abstinence/relapse attitudes, attitudes and use of adjunct strategies, and other smoking behaviors for adolescent smokers.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents presenting for regular well or sick visits at their pediatrician's office.
* Must live in a home or apartment with access to a telephone and mailing address.
* Must be able to speak English.
* Must be able and willing to give informed consent (if 18 years of age or older) or assent (if 14-17 years of age).
* In addition: parents/legal guardians of minors must be able and willing to give informed consent either in person or by phone in cases where the teen presents for care without a parent/legal guardian.

Exclusion Criteria:

* Adolescents who fall outside of the age range specified above.
* Unable to speak English.
* Do not have access to a telephone and/or mailing address.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10967 (Actual)
Dates: Start 2011-05; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in self-reported smoking status since baseline. | 4-6 weeks after initial doctor's visit, 6 months after initial doctors' visit, 12 months after initial doctor's visit.
  Via phone interview, adolescents will be asked to report their current smoking status, any quit-attempts, success of those quit-attempts, abstinence from tobacco products, and use of adjunct resources in the time since their initial doctor's visit.

SECONDARY OUTCOMES:
Adolescent-report of clinician visit. | 4-6 weeks after initial doctor visit
  In a phone interview, adolescents will be asked to report on the screenings, counseling, and referral to any cessation adjuncts that occured during their doctor visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D. Klein, MD, MPH, Principal Investigator — University of Illinois at Chicago and the American Academy of Pediatrics Julius B Richmond Center
Locations (1):
- American Academy of Pediatrics, Elk Grove Village, Illinois, United States

REFERENCES:
- [Derived] Klein JD, Gorzkowski J, Resnick EA, Harris D, Kaseeska K, Pbert L, Prokorov A, Wang T, Davis J, Gotlieb E, Wasserman R. Delivery and Impact of a Motivational Intervention for Smoking Cessation: A PROS Study. Pediatrics. 2020 Oct;146(4):e20200644. doi: 10.1542/peds.2020-0644. PMID 32989082